CLINICAL TRIAL: NCT05864339
Title: Efficacy of a Designed Empathy Course During Smoking Cessation Counseling Training for Nursing Students: A Randomized Controlled Trial
Brief Title: Efficacy of a Designed Empathy Course
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Derek Yee-Tak Cheung, Principal Investigator, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Empathy course protocol-v1
Record Dates: First submitted 2023-04-24; First posted 2023-05-18 (Actual); Last update posted 2023-05-18 (Actual); Status verified 2023-05

CONDITIONS: Smoking Cessation; Nursing Education
Keywords: Empathy; Nursing students; Nurse; Smoking cessation counseling; training
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Intervention Model Description: This study was designed based on Kolb's Experiential Learning Theory (ELT). This study is a 2-arm, randomized controlled trial (RCT) (allocation ratio 1:1), by comparing the empathy, self-efficacy, skill, attitude, and practice between master nursing students who participated in the designed empathy tutorial (viewing videos of four smokers' real-life scenarios, reading four smokers cases text materials, and drawing Health Empathy Map) (intervention group) and those who participated in a conventional tutorial (viewing videos of four smokers' real-life scenarios, reading four smokers cases text materials) (control group).
Who Masked: Participant
Masking Description: Participants will not know if they are given the the conventional tutorials or the newly designed empathy tutorials.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- A designed empathy tutorial during the SCC course (Intervention group) (Experimental): Students who participated in the designed empathy tutorial (viewing videos of four smokers' real-life scenarios, reading four smokers cases text materials, and drawing Health Empathy Map). Students will demonstrate a quit plan by role-playing and will attend focus group interviews during the wrap-up session.
  Interventions: Behavioral: A designed empathy intervention
- Smoking cessation counseling tutorial (Control group) (Active Comparator): Students will watch videos of four smokers' real-life scenarios, and read four smokers' case text materials. Students will demonstrate a quit plan by role-playing and will attend focus group interviews during the wrap-up session.
  Interventions: Behavioral: Smoking cessation counseling tutorial

INTERVENTIONS:
Behavioral: A designed empathy intervention — Students watch 4 smokers' videos, read the textual materials, fill out the HEMs and discuss a quit counseling plan for an assigned smoker using the 5As counseling skilll.
  Arms: A designed empathy tutorial during the SCC course (Intervention group)
Behavioral: Smoking cessation counseling tutorial — Students watch 4 smokers' videos, read the textual materials, and discuss a quit counseling plan for an assigned smoker using the 5As counseling skill.
  Arms: Smoking cessation counseling tutorial (Control group)

SUMMARY:
This proposed study aims to develop a designed empathy course intervention during the smoking cessation counseling (SCC) training for master nursing students at the University of Hong Kong.

The objectives are:

1. To increase master nursing students' empathy towards smokers.
2. To increase master nursing students' self-efficacy towards SCC.
3. To improve master nursing students' attitude towards SCC;
4. To increase master nursing students' use of 5As counseling skill(Ask, Advise, Assess, Assist, and Arrange) during their practice.

DETAILED DESCRIPTION:
1. Background:

   This proposed study was designed based on Kolb's Experiential Learning Theory (ELT). Kolb defined that learning requires the acquisition of abstract concepts that can then be applied flexibly in a wide range of situations. He created the experiential learning cycle in 1974, the four-stage model views learning as an integrated process. All four stages are mutually supportive because Kolb believes that effective learning is a cyclic process that involves experiencing, reflecting, thinking, and acting. The model for experiential learning theory portrays two dialectically related modes of grasping experience (concrete experience and abstract conceptualization) and two dialectically related modes of transforming experience (reflective observation and active experimentation), which help learners transform their experience into knowledge. Each of these stages acts as a foundation for the next stage.
2. Study design:

   This proposed study is a 2-arm, randomized controlled trial (RCT) (allocation ratio 1:1), by comparing the empathy, self-efficacy, attitude, and practice between master nursing students of two groups who participated in the designed empathy tutorial.
3. Subjects:

   The study targets to recruit students of Master of Nursing who are taking the course "Tobacco Dependency Nursing Intervention and Management (NURS8205)" in the spring semester, of 2023.
4. Procedures of teaching intervention:

   1. Students in both groups will watch the a smoker's video during the empathy course and fill out the Comprehensive State Empathy Scale based on their feeling towards the smoker in the video.
   2. The tutor will present slides about the importance of empathy and empathy skills in the SCC (the intervention group) and instruct students on how to fill out the Health Empathy Map(HEM) ( only for the intervention group). But students in the control group will receive the presentation about 5As counseling skill and do not be instructed on how to fill out the HEM.
   3. Students of both groups will be further allocated to 8 small groups with 3~5 participants. During the break-out session, students will watch 4 smokers' cases (A-D) via videos and textual materials. Each student fills out 4 HEMs for 4 smokers (the intervention group). Then, each small group in both groups has to discuss and prepare a quit plan for an assigned smoker using the 5As and will present by role play.
   4. Each small group (both groups) will recommend two students to demonstrate the smoking cessation counseling plan using the 5As , one student will play the "nurse" role, and the other student will play the "smoker" role. Each small group has 10 minutes to present, the tutor and other students can comment and feedback after each small group's presentation.
   5. After all presentations of the 8 small groups, the tutor will organize a focus group interview and instruct the students to complete the post-questionnaire at the end of the tutorial. Focus groups interview will be audio recorded while a research assistant served as a scribe.
5. Sample size calculate Sample size will be determined based on a G*Power analysis, using the t-test, to measure the difference between two independent means (two groups) to achieve a medium effect size of 0.8, A minimum sample size of 54 nursing students will be needed to achieve a power of 70% at 0.05 level of two-sided significance. To reach a meaningful result from the analysis of data, we added a buffer of 6 additional students (N = 60) to ensure the validity and robustness of the results.
6. Randomization and blinding The computer random number generator "Research Randomizer" will be used in the sequence generation process to generate a random sample using the block randomization technique. The single-blinding technique will be used to conceal the allocation. Participants will not know if they are given the conventional tutorials or the newly designed empathy tutorials.
7. Consent Students will receive an invitation email from the primary investigator and complete informed consent before the empathy course.
8. Statistical analysis Data will be entered into SPSS for Windows (version 20) for analysis. Descriptive statistics including frequency, percentage, and mean will be used to summarize the outcomes and other variables. By intention-to-treat analysis, participants who are lost or refuse the follow-up will be treated as having no change in the training outcomes. Chi-square tests and t-tests will be used to compare the outcomes between intervention and control groups. The effect size, Cohen's d, of the standardized mean of the pre-post differences will be computed, with and without adjustment for baseline characteristics. Linear mixed models which allow for multiple observations between subjects and account for the clustering of data within subjects will be used to assess the intervention effect on empathy, self-efficacy, attitude, and practice. Both the main effect (group allocation) and interaction effect (group X time) will be analyzed. To integrate and complement the obtained results, a qualitative analysis of the HEMs and focus group interview were performed using the content analysis technique, categorical modality, which is based on the decoding of a text into several elements that are then classified and form thematic groups that help to understand and describe the content of the messages.

ELIGIBILITY:
Inclusion Criteria:

* Master nursing students (1-2 years)
* Students are able to read, understand, and write in both English and Cantonese
* Students are willing to participate in this study and sign the informed consent.

Exclusion Criteria:

* Students who have taken any empathy courses in the past 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-25 (Estimated); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
The changes of empathy towards smokers | Change from before the empathy course and immediately after the empathy course (at the same day).
  The Comprehensive State Empathy Scale will be used to evaluate the master nursing students' empathy towards smokers. This scale has 30 items, each item is scored using a five-point Likert scale with response ranges from 1 (completely untrue) to 5 (completely true), with higher scores reflecting higher empathy levels, with the total scores ranging from 30 to 150 points.The higher score means the higher empathy.
The changes of self-efficacy towards smoking cessation counseling | Change from before the tutorial, after the tutorial and 2-month follow up.
  The sub-scale Self-efficacy of the Providers Smoking Cessation Training Evaluation will be used to assess the students' self-efficacy towards smoking cessation counseling. The total score ranges from 13 to 65 points, the higher score means the higher self-efficacy.

SECONDARY OUTCOMES:
The changes of students' attitude towards smoking cessation counseling | Change from before the tutorial, after the tutorial and 2-month follow up.
  The attitude sub-scale of The Providers Smoking Cessation Training Evaluation will be used to assess the students' attitude towards smoking cessation counseling.The total score ranges from 8 to 40 points, the higher score means the higher attitude.
The scores of students' 5As smoking cessation counseling skill | 2 weeks after the this entire course.
  The scores of the students' practical examination will be used to evaluate 5As smoking cessation counseling skill level that they have acquired.The total score ranges from 0 to 100 points, the higher score means the higher 5As skill.
The changes of students' practical behavior of smoking cessation counseling skill during their clinical workplace.The total score ranges from 8 to 40 points, the higher score means the higher attitude. | Change from before the tutorial at 2-month follow up.
  The behavior sub-scale of The Providers Smoking Cessation Training Evaluation will be used to assess the students' practical behavior of smoking cessation counseling.The total score ranges from 19 to 95 points, the higher score means the higher practical behavior.
The scores of students' satisfaction with the designed tutorial | Immediately after the empathy course.
  The 'Satisfaction' sub-scale from the Student Satisfaction and Self-Confidence in Learning Simulation will be revised to measure nursing students' satisfaction with the designed tutorial.The total score ranges from 5 to 25 points, the higher score means the higher satisfaction.
Qualitative measures | The wrap-up session during the empathy tutorial.
  Students will attend a focus group interview during the wrap-up session, and the following questions will be discussed: a)What are your personal experiences towards smokers in those videos? b)What comes to you mind when the smokers have quitting barriers in the videos. c)Do you think nurses should show empathy to smokers during the counseling? Why or why not ? d)What factors would affect your empathy towards smokers? e)What are some of the things nurses do when they show empathy towards smokers during the counseling? f)Do you think empathy levels in someone can be changed? Or is it inborn, meaning it cannot be taught. g)Please share you attitude, self-efficacy, and practice towards help smokers patients to quit after this training. h)Before ending the session, any more to you would like to share with us, about the tutorial or any others?
Qualitative contents of the Health Empathy Map | At the end of the 2-month trial period.
  The content analysis technique will be used to analysis the sentences on the Health Empathy Map that written by students.

CONTACTS AND LOCATIONS:
Overall Officials: Derek Yee Tak Cheung, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Research data and documentation will be available upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for 10 years.

REFERENCES:
- [Result] Bas-Sarmiento P, Fernandez-Gutierrez M, Baena-Banos M, Romero-Sanchez JM. Efficacy of empathy training in nursing students: A quasi-experimental study. Nurse Educ Today. 2017 Dec;59:59-65. doi: 10.1016/j.nedt.2017.08.012. Epub 2017 Sep 8. PMID 28945994
- [Result] Batt-Rawden SA, Chisolm MS, Anton B, Flickinger TE. Teaching empathy to medical students: an updated, systematic review. Acad Med. 2013 Aug;88(8):1171-7. doi: 10.1097/ACM.0b013e318299f3e3. PMID 23807099
- [Result] Cheung YTD, Chan CHH, Ho KS, Tang C, Lau CWH, Li WHC, Wang MP, Lam TH. Effectiveness of nicotine replacement therapy sample at outdoor smoking hotspots for initiating quit attempts and use of smoking cessation services: a protocol for a cluster randomised controlled trial. BMJ Open. 2020 Apr 7;10(4):e036339. doi: 10.1136/bmjopen-2019-036339. PMID 32269028
- [Result] Chun CK, Wong FK, Wang SL, Chen W. Examining advanced nursing practice in Hong Kong and Guangzhou. Int J Nurs Sci. 2021 Mar 5;8(2):190-198. doi: 10.1016/j.ijnss.2021.03.001. eCollection 2021 Apr 10. PMID 33997133
- [Result] Duaso MJ, Bakhshi S, Mujika A, Purssell E, While AE. Nurses' smoking habits and their professional smoking cessation practices. A systematic review and meta-analysis. Int J Nurs Stud. 2017 Feb;67:3-11. doi: 10.1016/j.ijnurstu.2016.10.011. Epub 2016 Nov 2. PMID 27880873
- [Result] Gholamzadeh S, Khastavaneh M, Khademian Z, Ghadakpour S. The effects of empathy skills training on nursing students' empathy and attitudes toward elderly people. BMC Med Educ. 2018 Aug 15;18(1):198. doi: 10.1186/s12909-018-1297-9. PMID 30111312
- [Result] Hasan SI, Mohd Hairi F, Ahmad Tajuddin NA, Amer Nordin AS. Empowering healthcare providers through smoking cessation training in Malaysia: a preintervention and postintervention evaluation on the improvement of knowledge, attitude and self-efficacy. BMJ Open. 2019 Sep 27;9(9):e030670. doi: 10.1136/bmjopen-2019-030670. PMID 31562154
- [Result] Hasan SI, Mohd Hairi F, Amer Nordin AS, Danaee M. Development and Validation of an Evaluation Tool to Measure the Effectiveness of a Smoking Cessation Training among Healthcare Providers in Malaysia: The Providers' Smoking Cessation Training Evaluation (ProSCiTE). Int J Environ Res Public Health. 2019 Nov 5;16(21):4297. doi: 10.3390/ijerph16214297. PMID 31694286
- [Result] Levett-Jones T, Cant R, Lapkin S. A systematic review of the effectiveness of empathy education for undergraduate nursing students. Nurse Educ Today. 2019 Apr;75:80-94. doi: 10.1016/j.nedt.2019.01.006. Epub 2019 Jan 26. PMID 30739841
- [Result] Luo YF, Chen LC, Yang SC, Hong S. Knowledge, Attitude, and Practice (KAP) toward COVID-19 Pandemic among the Public in Taiwan: A Cross-Sectional Study. Int J Environ Res Public Health. 2022 Feb 27;19(5):2784. doi: 10.3390/ijerph19052784. PMID 35270491
- [Result] Patterson J, Duke G, Stocks E, Hermanns M. Simulation to Enhance Empathy of Nursing Students Toward Patients With Alcohol Use Disorder: A Mixed-Methods Study. Nurse Educ. 2020 Nov/Dec;45(6):331-335. doi: 10.1097/NNE.0000000000000804. PMID 31972845
- [Result] Harizi C, El-Awa F, Ghedira H, Audera-Lopez C, Fakhfakh R. Implementation of the WHO Framework Convention on Tobacco Control in Tunisia: Progress and challenges. Tob Prev Cessat. 2020 Dec 22;6:72. doi: 10.18332/tpc/130476. eCollection 2020. PMID 33426382
- [Derived] Zhang G, Luk TT, Lam VSF, Zhao S, Yip AON, Wang MP, Chan SSC, Cheung YTD. Effectiveness of a theory-based empathy enhancement in increasing Master of Nursing students' empathy and practice of smoking cessation intervention: A randomized controlled trial. Nurse Educ Pract. 2025 Aug;87:104483. doi: 10.1016/j.nepr.2025.104483. Epub 2025 Jul 23. PMID 40714657